CLINICAL TRIAL: NCT04838626
Title: Phase II/III Study for Evaluation of the Diagnostic Performance of [18F]CTT1057 PET Imaging for the Detection of PSMA Positive Tumors Using Histopathology as a Standard of Truth
Brief Title: Study of Diagnostic Performance of [18F]CTT1057 for PSMA-positive Tumors Detection
Acronym: GuideView
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CAAA405A12302; 2020-003958-67 (EudraCT Number)
Record Dates: First submitted 2021-04-07; First posted 2021-04-09 (Actual); Results first posted 2024-12-18 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Prostatic Neoplasms; Prostate Cancer
Keywords: [18F]CTT1057; Positron Emission Tomography/Computerized Tomography; PET/CT; Radioligand; Imaging; Primary Staging; PS; Standard of Truth; SoT; Prostate Cancer; PCa
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: All participants will receive [18F]CTT1057 for PET/CT scan imaging, and surgery will be performed up to 6 weeks after [18F]CTT1057 PET for pathology assessment of the tissue specimens.
  Additional pharmacokinetics (PK) assessments will be performed on the date of imaging in a subset of approximately 10 patients at the same site.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PET/CT imaging with [18F]CTT1057 (Experimental): All eligible participants will be enrolled to receive [18F]CTT1057 imaging agent on Day 1 and have PET/CT scan
  Interventions: Drug: [18F]CTT1057

INTERVENTIONS:
Drug: [18F]CTT1057 — PET/CT imaging with [18F]CTT1057
  Other Names: Single intravenous dose of approximately 370 Mega-Becquerel (MBq) and subsequent PET/CT scan

SUMMARY:
The purpose of this study was to evaluate the diagnostic performance of [18F]CTT1057 as a PET imaging agent for detection and localization of PSMA positive tumors using histopathology as Standard of Truth (SoT). Tissue specimens from both the primary tumor and pelvic lymph nodes dissected during surgery from patients with newly-diagnosed high-risk prostate cancer (PCa) were used for the histopathology assessments.

DETAILED DESCRIPTION:
This was a multi-center, single-arm, open-label prospective study to evaluate the diagnostic performance of vidoflufolastat (18F) as a positron emission tomography (PET) imaging agent for detection and localization of prostate specific membrane antigen (PSMA) positive tumors, using histopathology as standard of truth (SoT). in newly diagnosed high-risk prostate cancer (PCa) patients.

A total of 195 participants were enrolled to ensure that at least 156 participants were evaluable for the co-primary endpoints. Surgery was performed after vidoflufolastat (18F) positron emission tomography/computerized tomography (PET/CT) scan.

The co-primary endpoints of patient-level sensitivity and region-level specificity were assessed by comparing the central reading results of the vidoflufolastat (18F) PET/CT scan to the local histopathology results in the dissected tissue specimens, i.e. both the primary tumor and the dissected Pelvic Lymph Nodes (PLNs).

ELIGIBILITY:
Inclusion Criteria:

* Untreated high risk biopsy-proven PCa patients according to D'Amico classification (Stage ≥ T2c or PSA level >20ng/ml or Gleason score ≥8) (D'Amico et al 1998)
* Scheduled or planned radical prostatectomy and extended pelvic lymph node resection up to 6 weeks after the investigational PET/CT scan followed by histopathology assessment
* ECOG performance status 0-2
* Signed informed consent must be obtained prior to participation in the study
* Participants must be adults ≥ 18 years of age

Exclusion Criteria:

* Inability to complete the needed investigational and standard-of-care imaging examinations due to any reason (severe claustrophobia, inability to lie still for the entire imaging time, etc.)
* Any additional medical condition, serious intercurrent illness, concomitant cancer or other extenuating circumstance that, in the opinion of the Investigator, would indicate a significant risk to safety or impair study participation, including, but not limited to, current severe urinary incontinence, hydronephrosis, severe voiding dysfunction, need of indwelling/condom catheters, New York Heart Association class III or IV congestive heart failure, history of congenital prolonged QT syndrome, uncontrolled infection, active hepatitis B or C, and COVID-19.
* Known allergy, hypersensitivity, or intolerance to [18F]CTT1057
* Prior and current use of PSMA targeted therapies
* Prior and current treatment with any ADT (first or second generation), including LHRH analogues (agonists or antagonists)
* Any 5-alpha reductase inhibitors within 30 days before screening
* Patients with small cell or neuroendocrine PCa in more than 50% of biopsy tissue
* Patients with incidental PCa after transurethral resection
* Use of other investigational drugs within 30 days before screening

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2021-09-07 (Actual); Primary Completion 2023-11-24 (Actual); Study Completion 2023-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (13):
- Explorer Molecular Imaging center, Sacramento, California, United States
- France (4):
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Nîmes
  - Novartis Investigative Site, Pierre-Bénite
  - Novartis Investigative Site, Toulouse
- Italy (3):
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
- Spain (3):
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Barcelona
- Switzerland (2):
  - Novartis Investigative Site, Bellinzona
  - Novartis Investigative Site, Geneva

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://clinicalstudydatarequest.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 195 patients were enrolled. 184 participants received vidoflufolastat (18F) and 184 underwent PET/CT. 173 patients completed the study and 184 patients completed treatment.
Groups:
- PET/CT Imaging With Vidoflufolastat (18F).: Single intravenous dose of approximately 370 Mega-Becquerel (MBq) on Day 1 and subsequent PET/CT scan
Period: Overall Study
Arm/Group | PET/CT Imaging With Vidoflufolastat (18F).
Started | 195
Participants Who Received Vidoflufolastat (18F) and Underwent PET/CT | 184
Completed | 173
Not Completed | 22
Not completed — Adverse Event | 2
Not completed — Physician Decision | 6
Not completed — Protocol Violation | 3
Not completed — Withdrawal by Subject | 9
Not completed — Technical Problems | 2

BASELINE CHARACTERISTICS:
Arm/Group | PET/CT Imaging With Vidoflufolastat (18F).
Number analyzed (Participants) | 195
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.5 (6.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 195
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 56
  Not Hispanic or Latino | 122
  Unknown or Not Reported | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 192
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Patient-level Sensitivity of Vidoflufolastat (18F) - % Sensitivity
Description: Sensitivity of vidoflufolastat (18F) Positron Emission Tomography (PET) imaging, considering Prostate Specific Membrane Antigen (PSMA) positive patients as those who show at least one pathological vidoflufolastat (18F) uptake either in the primary tumor and/or metastatic Pelvic Lymph Node (PLN) regions, with anatomically localized correspondence with the Standard of Truth (SoT).
Time Frame: vidoflufolastat (18F)7 PET imaging acquired at Day 1 assessed against histopathology as Standard of Truth (SoT) obtained during surgery within 6 weeks from vidoflufolastat (18F) scan
Population: The Efficacy Analysis Set (EFF) included all enrolled participants who received the dose of investigational treatment (i.e. vidoflufolastat (18F)), had both an evaluable vidoflufolastat (18F) PET/CT scan and histopathology assessment, and had not received any prohibited systemic antineoplastic therapy before the completion of PET/CT and surgery.
Measure: Number (95% Confidence Interval); unit: % Sensitivity
Groups:
- Central Reader 1: Central Reading Center 1
- Central Reader 2: Central Reading Center 2
- Central Reader 3: Central Reading Center 3
Arm/Group | Central Reader 1 | Central Reader 2 | Central Reader 3
Number analyzed (Participants) | 172 | 172 | 172
% Sensitivity | 86.8 [80.74 to 91.56] | 90.0 [84.47 to 94.07] | 86.9 [80.85 to 91.61]

2. Primary Outcome: Region-level Specificity of Vidoflufolastat (18F) - % Specificity
Description: Specificity of vidoflufolastat (18F) PET imaging, defined as proportion of PLN regions that test negative for lymph nodes on vidoflufolastat (18F) among those that are lymph node negative on the SoT.
Time Frame: vidoflufolastat (18F) PET imaging acquired at Day 1 assessed against histopathology as Standard of Truth (SoT) obtained during surgery within 6 weeks from vidoflufolastat (18F) scan
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: % Specificity
Arm/Group | Central Reader 1 | Central Reader 2 | Central Reader 3
Number analyzed (Participants) | 172 | 172 | 172
% Specificity | 97.1 [92.74 to 99.20] | 97.1 [92.74 to 99.20] | 97.1 [92.74 to 99.20]

3. Secondary Outcome: Patient-level Specificity of Vidoflufolastat (18F) - % Specificity
Description: Specificity of vidoflufolastat (18F) PET imaging, considering PSMA negative patients as those who do not show any pathological vidoflufolastat (18F) uptake either in the primary tumor or PLNs and will be confirmed not having primary tumor or metastatic PLNs with the SoT
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: % Specificity
Arm/Group | Central Reader 1 | Central Reader 2 | Central Reader 3
Number analyzed (Participants) | 172 | 172 | 172
% Specificity | 20.0 [0.51 to 71.64] | 0.0 [0.0 to 84.19] | 25.0 [0.63 to 80.59]

4. Secondary Outcome: Patient-level Positive Predictive Value of Vidoflufolastat (18F)
Description: Proportion of patients who are both vidoflufolastat (18F) and SoT positive (true positives (TP) among those who test positive on vidoflufolastat (18F) (TP+ false positives (FP))
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: % Positive Predictive Value
Arm/Group | Central Reader 1 | Central Reader 2 | Central Reader 3
Number analyzed (Participants) | 172 | 172 | 172
% Positive Predictive Value | 97.3 [93.27 to 99.26] | 98.7 [95.42 to 99.84] | 98.0 [94.23 to 99.58]

5. Secondary Outcome: Patient-level Negative Predictive Value of Vidoflufolastat (18F)
Description: Proportion of patients who are both vidoflufolastat (18F) and SoT negative (true negatives (TN)) among those who test negative on vidoflufolastat (18F) (TN+ false negatives (FN))
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: % Negative Predictive Value
Arm/Group | Central Reader 1 | Central Reader 2 | Central Reader 3
Number analyzed (Participants) | 172 | 172 | 172
% Negative Predictive Value | 4.3 [0.11 to 21.95] | 0.0 [0.0 to 19.51] | 4.3 [0.11 to 21.95]

6. Secondary Outcome: Patient-level Accuracy of Vidoflufolastat (18F)
Description: Proportion of patients that are SoT and vidoflufolastat (18F) positive (TP) and negative (TN) among all patients in Efficacy Analysis Set (EFF) (TP+TN+FP+FN)
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: % Accuracy
Arm/Group | Central Reader 1 | Central Reader 2 | Central Reader 3
Number analyzed (Participants) | 172 | 172 | 172
% Accuracy | 84.9 [78.64 to 89.88] | 89.0 [83.29 to 93.22] | 85.5 [79.30 to 90.37]

7. Secondary Outcome: Region-level Sensitivity of Vidoflufolastat (18F) - % Sensitivity
Description: Proportion of PLN regions that test positive on both vidoflufolastat (18F) and SoT (TP) among those that are SoT positive (TP+FN)
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: % Sensitivity
Arm/Group | Central Reader 1 | Central Reader 2 | Central Reader 3
Number analyzed (Participants) | 172 | 172 | 172
% Sensitivity | 20.6 [8.70 to 37.90] | 20.6 [8.70 to 37.90] | 23.5 [10.75 to 41.17]

8. Secondary Outcome: Region-level Positive Predictive Value of Vidoflufolastat (18F)
Description: Proportion of Pelvic Lymph Node (PLN) regions that are Standard of Truth (SoT) and vidoflufolastat (18F) positive (TP) among those regions that test positive on vidoflufolastat (18F) (TP+False Positive (FP))
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: % Positive Predictive Value
Arm/Group | Central Reader 1 | Central Reader 2 | Central Reader 3
Number analyzed (Participants) | 172 | 172 | 172
% Positive Predictive Value | 63.6 [30.79 to 89.07] | 63.6 [30.79 to 89.07] | 66.7 [34.89 to 90.08]

9. Secondary Outcome: Region-level Negative Predictive Value of Vidoflufolastat (18F)
Description: Proportion of PLN regions that are SoT and vidoflufolastat (18F) negative (TN) among those regions that test negative on vidoflufolastat (18F) (TN+FN)
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: % Negative Predictive Value
Arm/Group | Central Reader 1 | Central Reader 2 | Central Reader 3
Number analyzed (Participants) | 172 | 172 | 172
% Negative Predictive Value | 83.2 [76.55 to 88.65] | 83.2 [76.55 to 88.65] | 83.8 [77.10 to 89.10]

10. Secondary Outcome: Region-level Accuracy of Vidoflufolastat (18F)
Description: Proportion of PLN regions that are SoT and vidoflufolastat (18F) positive (TP) and negative (TN) among all PLN regions assessed vidoflufolastat (18F)(TP+TN+FP+FN)
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: % Accuracy
Arm/Group | Central Reader 1 | Central Reader 2 | Central Reader 3
Number analyzed (Participants) | 172 | 172 | 172
% Accuracy | 82.0 [75.40 to 87.41] | 82.0 [75.40 to 87.41] | 82.6 [76.05 to 87.91]

11. Secondary Outcome: Region-level Sensitivity of Vidoflufolastat (18F) Scan With Standard of Truth Excluding Pelvic Lymph Node (PLN) Metastasis < 2 mm
Description: Sensitivity of vidoflufolastat (18F) PET imaging in the PLN region, excluding from the analysis those lymph nodes showing metastasis <2mm (micro-metastasis)
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: % Sensitivity
Arm/Group | Central Reader 1 | Central Reader 2 | Central Reader 3
Number analyzed (Participants) | 172 | 172 | 172
% Sensitivity | 26.9 [11.57 to 47.79] | 26.9 [11.57 to 47.79] | 30.8 [14.33 to 51.79]

12. Secondary Outcome: Detection of Distant Metastasis of Vidoflufolastat (18F) Scan - Participants With at Least One Distant Metastatic Lesion (%)
Description: Number of distant metastasis identified at PET/CT scan in all patients, and percentage of patients with at least one distant metastatic lesion (extra-PLN, visceral or skeletal)identified by PET scan in all patients with an evaluable vidoflufolastat (18F) PET/CT scan.
Time Frame: as for outcome 2
Population: Safety set - all treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | Central Reader 1 | Central Reader 2 | Central Reader 3
Number analyzed (Participants) | 184 | 184 | 184
Participants | 6 | 9 | 10

13. Secondary Outcome: Overview of Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence (e.g. any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a subject or clinical investigation subject
Time Frame: Adverse Events are reported from the single dose of study treatment administration until 14 days afterwards, for a maximum time frame of approx. 14 days.
Population: Safety set - all treated patients
Measure: Count of Participants; unit: Participants
Groups:
- PET/CT Imaging With Vidoflufolastat (18F).: Study participants were injected intravenously with approximately 370 MBq (range 266 - 407 MBq) of vidoflufolastat (18F).
Arm/Group | PET/CT Imaging With Vidoflufolastat (18F).
Number analyzed (Participants) | 184
Participants
  Adverse events | 24
  Treatment-related Adverse events | 1
  Serious adverse events | 2
  Serious adverse events Treatment-related | 0
  Fatal serious adverse events | 0
  Fatal serious adverse events Treatment-related | 0
  Adverse events leading to dose adjustment / interruption | 0
  Adverse events requiring additional therapy | 5

14. Secondary Outcome: Vidoflufolastat (18F) Scan Inter-reader Variability - %
Description: Scan inter-reader variability is defined the agreement rate among reader determination of vidoflufolastat (18F) images.
Time Frame: as for outcome 2
Population: Safety set - all treated patients
Measure: Number (95% Confidence Interval); unit: % variability
Arm/Group | PET/CT Imaging With Vidoflufolastat (18F).
Number analyzed (Participants) | 184
% variability | 63.9 [55.52 to 72.20]

15. Secondary Outcome: Vidoflufolastat (18F) Scan Inter-reader Variability - Number of Scans Agreed
Description: Scan inter-reader variability is defined the agreement rate among reader determination of vidoflufolastat (18F) images.
Time Frame: as for outcome 2
Population: Safety set - all treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | PET/CT Imaging With Vidoflufolastat (18F).
Number analyzed (Participants) | 184
Participants
  Number of scans agreed by all three readers | 163
  Number of scans agreed by two readers | 21

16. Secondary Outcome: Vidoflufolastat (18F) Scan Intra-reader Variability
Description: Scan intra-reader variability is defined as the within-reader agreement rate of vidoflufolastat (18F) images.
Time Frame: as for outcome 2
Population: Safety set - all treated patients with a valid measurement.
  For this outcome measure, scans for a subset of 20 patients were read by each reader at 2 different time points.
Measure: Number (95% Confidence Interval); unit: variability (%)
Groups:
- Central Reader 1: Central Reader 1
- Central Reader 2: Central Reader 2
- Central Reader 3: Central Reader 3
Arm/Group | Central Reader 1 | Central Reader 2 | Central Reader 3
Number analyzed (Participants) | 20 | 20 | 20
variability (%) | 100 [100 to 100] | 100 [100 to 100] | 89.4 [69.0 to 100]

17. Secondary Outcome: Observed Maximum Blood Concentration (Cmax) of Vidoflufolastat (18F)
Time Frame: Day 1 (0, 0-5, 15, 30, 60, 120, 180-240, 300 minutes post injection)
Population: The Pharmacokinetic analysis set (PAS) included all participants who received the investigational treatment (i.e. vidoflufolastat (18F)) with valid results for the outcome measure.
  For PK outcome measures, a subset of 10 patients maximum were analyzed.
Measure: Mean (Standard Deviation); unit: kBq/mL
Arm/Group | PET/CT Imaging With Vidoflufolastat (18F).
Number analyzed (Participants) | 10
kBq/mL | 49.0 (19.2)

18. Secondary Outcome: Time of Maximum Observed Blood Concentration Occurrence (Tmax) of Vidoflufolastat (18F)
Time Frame: Day 1 (0, 0-5, 15, 30, 60, 120, 180-240, 300 minutes post injection)
Population: as for outcome 17
Measure: Median (Full Range); unit: Hours
Arm/Group | PET/CT Imaging With Vidoflufolastat (18F).
Number analyzed (Participants) | 10
Hours | 0.0333 [0.0167 to 0.0833]

19. Secondary Outcome: Area Under the Vidoflufolastat (18F) Concentration-time Curve From Time Zero to the Time of Last Quantifiable Concentration (AUClast)
Time Frame: Day 1 (0, 0-5, 15, 30, 60, 120, 180-240, 300 minutes post injection)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: h*kBq/mL
Arm/Group | PET/CT Imaging With Vidoflufolastat (18F).
Number analyzed (Participants) | 10
h*kBq/mL | 47.9 (11.9)

20. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero (Pre-dose) Extrapolated to Infinite Time (AUCinf) of Vidoflufolastat (18F)
Time Frame: Day 1 (0, 0-5, 15, 30, 60, 120, 180-240, 300 minutes post infusion)
Population: The Pharmacokinetic analysis set (PAS) included all participants who received the investigational treatment (i.e. vidoflufolastat (18F)) with valid results for the outcome measure.
  For PK outcome measures, a subset of 10 patients maximum were analyzed. For this parameter, results for only 1 pt were evaluable.
Measure: Mean (Standard Deviation); unit: h*kBq/mL
Arm/Group | PET/CT Imaging With Vidoflufolastat (18F).
Number analyzed (Participants) | 1
h*kBq/mL | 50.0 (NA) — not applicable when n = 1

21. Secondary Outcome: Half-Life Lambda z of Vidoflufolastat (18F)
Time Frame: Day 1 (0, 0-5, 15, 30, 60, 120, 180-240, 300 minutes post injection)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: h
Arm/Group | PET/CT Imaging With Vidoflufolastat (18F).
Number analyzed (Participants) | 1
h | 1.34 (NA) — not applicable when n = 1

22. Secondary Outcome: Volume of Distribution During the Terminal Phase Following Intravenous Elimination (Vz) of Vidoflufolastat (18F)
Time Frame: Day 1 (0, 0-5, 15, 30, 60, 120, 180-240, 300 minutes post injection)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: L
Arm/Group | PET/CT Imaging With Vidoflufolastat (18F).
Number analyzed (Participants) | 1
L | 14.9 (NA) — not applicable when n = 1

23. Secondary Outcome: Urinary Excretion of Radioactivity Expressed as a Percentage of Injected Activity (%IA) of Vidoflufolastat (18F)
Time Frame: Day 1 (pre-injection/0 hour, 0 hour (injection) - T (image acquisition starting time), T (image acquisition starting time) to 3 hours, 3 hours to 5 hours post imaging)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: %IA
Arm/Group | PET/CT Imaging With Vidoflufolastat (18F).
Number analyzed (Participants) | 10
%IA
  0 HRS INJECTION/PRE-INJECTION | 0.000821 (0.00120)
  0 HRS (INJECTION) - T (IMAGE ACQUISITION STARTING TIME) | 15.8 (11.9)
  IMAGE ACQUISITION STARTING TIME T - 3 H | 11.9 (8.30)
  3 H - 5 H | 10.5 (8.06)

24. Secondary Outcome: Total Systemic Clearance for Intravenous Administration (CL) of Vidoflufolastat (18F)
Time Frame: Day 1 (0, 0-5, 15, 30, 60, 120, 180-240, 300 minutes post injection)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | PET/CT Imaging With Vidoflufolastat (18F).
Number analyzed (Participants) | 1
L/h | 7.70 (NA) — not applicable when n = 1

ADVERSE EVENTS:
Time Frame: Adverse Events are reported from the single dose of study treatment administration until 14 days afterwards, for a maximum time frame of approx. 14 days.
Arm/Group | PET/CT Imaging With Vidoflufolastat (18F)
All-Cause Mortality (participants affected / at risk) | 0/184
Serious Adverse Events (participants affected / at risk) | 2/184
Other Adverse Events (participants affected / at risk) | 23/184
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PET/CT Imaging With Vidoflufolastat (18F) (N=184)
Myocardial ischaemia (Cardiac disorders) | 1
Sepsis syndrome (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PET/CT Imaging With Vidoflufolastat (18F) (N=184)
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Feeling hot (General disorders) | 1
Pyrexia (General disorders) | 1
COVID-19 (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Amylase increased (Investigations) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 2
Insomnia (Psychiatric disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Scrotal oedema (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 1
Hot flush (Vascular disorders) | 1
Hypertension (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-12-20): https://cdn.clinicaltrials.gov/large-docs/26/NCT04838626/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-26): https://cdn.clinicaltrials.gov/large-docs/26/NCT04838626/SAP_001.pdf